CLINICAL TRIAL: NCT00286000
Title: High Dose Simplified Folfiri in Advanced Colorectal Cancer: a Multicentre Phase II Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004/195
Record Dates: First submitted 2006-02-01; First posted 2006-02-02 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Advanced Colorectal Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Administration of high dose simplified folfiri

SUMMARY:
A multicentre phase II study to evaluate the results of high dose simplified folfiri in advanced colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven adenocarcinoma of the colon or rectum
* Documented progressive metastatic disease
* Patients who have at least one uni-dimensional measurable lesion by CT-scan or MRI according to response evaluation criteria in solid tumours (RECIST)
* WHO performance status of 0 or 1
* Adequate laboratory values of haematology, liverfunction and renal function
* No previous chemotherapy for metastatic colorectal cancer

Exclusion Criteria:

* Past or concurrent history of neoplasm other than colorectal adenocarcinoma, except curatively treated cancer free of disease for more than 10 years.
* Bowel obstruction or sub-obstruction. Crohn's disease, or ulcerative colitis.
* Other severe illness or medical condition such as unstable cardiac disease under treatment, myocardial infarction within 6 months before inclusion.
* Active uncontrolled infection
* Other concomitant anticancer agent

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106
Dates: Start 2004-06; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Response rate

SECONDARY OUTCOMES:
Resectability
Safety
TTP

CONTACTS AND LOCATIONS:
Overall Officials: Marc Peeters, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be